CLINICAL TRIAL: NCT05710718
Title: A Comparative Crossover Study on the Safety, Efficacy, and Patient Quality of Life Comparing PureWick™ System With an Established Comparator in the Home Setting for Incontinence Overnight
Brief Title: PureWick™ France and U.S. At-Home Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Collaborators: Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: UCC-8007
Record Dates: First submitted 2023-01-04; First posted 2023-02-02 (Actual); Results first posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-05

CONDITIONS: Nocturnal Enuresis
MeSH Terms: conditions — Nocturnal Enuresis

STUDY DESIGN:
Intervention Model Description: 1:1 Crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Treatment Sequence 1 (Other): The PureWick™ System is used for the first 4 weeks, followed by cross-over to the Hollister Female Urinary Pouch.
  Interventions: Device: PureWick™ System; Device: Hollister® Female Urinary Pouch External Collection Device
- Treatment Sequence 2 (Other): The Hollister Female Urinary Pouch is used for the first 4 weeks, followed by cross-over to the PureWick™ System.
  Interventions: Device: PureWick™ System; Device: Hollister® Female Urinary Pouch External Collection Device

INTERVENTIONS:
Device: PureWick™ System — The PureWick™ FEC is intended for non-invasive urine output management in female patients. The PureWick™ FEC is a flexible, contoured external catheter that is positioned against the area where urine exits the female body. The PureWick™ FEC is connected to the PureWick™ Urine Collection System (PUCS) via connector tubing. The PUCS uses suction (not felt by the user) to pull voided urine through the device, regardless of the urine flow rate. Urine continues through vinyl tubing until it reaches a collection canister, away from the body.
Device: Hollister® Female Urinary Pouch External Collection Device — The Hollister Female Urinary Pouch External Collection Device is intended to collect and contain urine for individuals with urinary incontinence. It is designed to be emptied and should be attached to a drainage bag. The FUP is made with hydrocolloid skin adhesive and polymer/copolymer plastics.

SUMMARY:
In this prospective, post-market, multi-site, open-label, crossover trial, women with urinary incontinence requiring the use of diapers (changes complets (French term)) at night will be 1:1 randomized to a treatment sequence using two devices (PureWick™ System and Hollister® Female Urinary Pouch External Collection Device) and followed for approximately 10 weeks through 2 treatment phases. The primary objectives are to evaluate safety (skin injury) and efficacy (capture rate). Safety will be assessed using the Draize Scale and efficacy will be measured based on daily urine capture rate.

DETAILED DESCRIPTION:
In this prospective, post-market, multi-site, open-label, crossover trial, women with urinary incontinence requiring the use of diapers (changes complets (French term)) at night will be 1:1 randomized to a treatment sequence using two devices (PureWick™ System and Hollister® Female Urinary Pouch External Collection Device) and followed for approximately 10 weeks through 2 treatment phases.

Approximately 30 female participants from 2 sites will be enrolled into the study. Those meeting eligibility criteria will be treated according to the treatment sequence assigned during randomization. Participants will view the standardized training video for the applicable product at the beginning of each treatment phase and have access to the Information for Use document (IFU) to review during each treatment phase. The total expected duration of subject participation is approximately 10 weeks. Participants will use the device assigned in treatment phase 1 overnight while sleeping for 4 weeks (28 days) before transitioning to the second assigned device in treatment phase 2. There will be a minimum washout period of 2 weeks (not to exceed 4 weeks) between treatment phases and a re-screening of eligibility criteria before the second phase. In both treatment phases, participants will independently place and remove the FEC (female external catheter) or FUP (Female Urinary Pouch) after standardized teaching is completed on the first day of the treatment phase.

The primary objectives are to evaluate safety (skin injury) and efficacy (capture rate). Safety will be assessed using the Draize Scale and efficacy will be measured based on daily urine capture rate. Health Care Providers (HCPs) will visit participants' homes daily to perform a skin assessment and collect urine measurements during the treatment phases. Participants will be withdrawn from the treatment phase if grade 4 is achieved in any category on the Draize skin irritation scale.

The secondary objectives are to assess quality of life, tolerability, comfort and ease of use. Quality of life and comfort and ease of use will be measured using self-reported changes in quality of life via the validated Nocturia Quality of Life (N-Qol) tool & the PROMIS Sleep Disturbance Short-form 4a survey, and subjective evaluation of the therapy via participant survey, respectively. Tolerability will be measured by number of days of actual use of both devices, and discontinuation rate attributed to the device's discomfort or inconvenience.

ELIGIBILITY:
Inclusion Criteria:

1. Adult Female Participants >18 years of age at the time of signing the informed consent.
2. Currently use diapers or equivalent at night for urine capture ("Change complet"(French term))
3. Willing to comply with all study procedures in the protocol
4. Provision of signed and dated informed consent form

Exclusion Criteria:

1. Has frequent episodes of bowel incontinence without a fecal management system in place; or
2. Has moderate to heavy menstruation and cannot use a tampon or menstrual cup; or
3. Has Urinary tract, vaginal or other chronic infections, active genital herpes; or
4. Has Urinary retention; or
5. Is agitated, combative, and/or uncooperative and may remove the external catheter or pouch; or
6. Has any wound, open lesion or irritation on the genitalia, perineum, or sacrum; or
7. Has any pre-existing neurological, psychiatric, or other condition that would confound quality of life assessment or would make it difficult to self-report on quality-of-life questionnaires in the opinion of the investigator; or
8. Is known to be pregnant at time of enrollment (for women of childbearing age); or
9. Any other condition that, in the opinion of the investigator, would preclude them from participating in the study.
10. Is under supervision of a legally authorized representative.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2023-10-31 (Actual); Primary Completion 2024-08-25 (Actual); Study Completion 2024-08-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Smiths Medical Center, Dunwoody, Georgia
  - Weill Cornell Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential subjects were identified and enrolled by the participating clinical research sites.
Pre-assignment Details: All enrolled participants were randomized to a treatment assignment; however, four (4) participants discontinued prior to starting treatment. The number of Started participants (13) represents those participants that were randomized and treated.
Groups:
- PureWick System, Then Hollister Female Urinary Pouch: The PureWick™ System is used for the first 4 weeks, followed by cross-over to the Hollister Female Urinary Pouch.
  PureWick™ System: The PureWick™ FEC is intended for non-invasive urine output management in female patients. The PureWick™ FEC is a flexible, contoured external catheter that is positioned against the area where urine exits the female body. The PureWick™ FEC is connected to the PureWick™ Urine Collection System (PUCS) via connector tubing. The PUCS uses suction (not felt by the user) to pull voided urine through the device, regardless of the urine flow rate. Urine continues through vinyl tubing until it reaches a collection canister, away from the body.
  Hollister® Female Urinary Pouch External Collection Device: The Hollister Female Urinary Pouch External Collection Device is intended to collect and contain urine for individuals with urinary incontinence. It is designed to be emptied and should be attached to a drainage bag. The FUP is made with hydrocolloid skin adhesive and polymer/copolymer plastics.
- Hollister Female Urinary Pouch, Then PureWick System: The Hollister Female Urinary Pouch is used for the first 4 weeks, followed by cross-over to the PureWick™ System.
  PureWick™ System: The PureWick™ FEC is intended for non-invasive urine output management in female patients. The PureWick™ FEC is a flexible, contoured external catheter that is positioned against the area where urine exits the female body. The PureWick™ FEC is connected to the PureWick™ Urine Collection System (PUCS) via connector tubing. The PUCS uses suction (not felt by the user) to pull voided urine through the device, regardless of the urine flow rate. Urine continues through vinyl tubing until it reaches a collection canister, away from the body.
  Hollister® Female Urinary Pouch External Collection Device: The Hollister Female Urinary Pouch External Collection Device is intended to collect and contain urine for individuals with urinary incontinence. It is designed to be emptied and should be attached to a drainage bag. The FUP is made with hydrocolloid skin adhesive and polymer/copolymer plastics.
Period: Overall Study
Arm/Group | PureWick System, Then Hollister Female Urinary Pouch | Hollister Female Urinary Pouch, Then PureWick System
Started | 6 | 7
Completed Treatment 1 | 5 | 1
Completed Treatment 2 | 1 | 4
Completed | 1 | 4
Not Completed | 5 | 3
Not completed — Withdrawal by Subject | 5 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants were randomized and treated.
Groups:
- PureWick, Then Hollister Female Urinary Pouch: The PureWick™ System is used for the first 4 weeks, followed by cross-over to the Hollister Female Urinary Pouch.
- Hollister Female Urinary Pouch, Then PureWick: The Hollister Female Urinary Pouch is used for the first 4 weeks, followed by cross-over to the PureWick™ System.
- Total: Total of all reporting groups
Arm/Group | PureWick, Then Hollister Female Urinary Pouch | Hollister Female Urinary Pouch, Then PureWick | Total
Number analyzed (Participants) | 6 | 7 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 5 | 6 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.3 (11.1) | 76.3 (18.0) | 75.3 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 7 | 12
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 7 | 10
  White | 3 | 0 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Daily Average Urine Capture Rate (Percentage)
Description: Capture rate following void (captured as % of urine captured by device and collected in canister, measured by weight).
  Prior to each nightly use, the weight of the empty urine collection canister and the weight of a dry absorbent pad are collected. Participants use the device overnight while sleeping with the absorbent pad underneath them. The next morning, the post-void weight of the urine collection canister and the post-void weight of the absorbent pad are collected.
  Capture rate is calculated as the weight of captured urine (post-void canister weight - pre-void canister weight) / total urine volume (captured urine (post-void canister weight - pre-void canister weight) + leaked urine (post-void pad weight - pre-void pad weight)) * 100.
  The primary efficacy endpoint of urine capture rate is derived by computing the mean of daily capture rate during each study phase.
Time Frame: Daily for 28 days during each treatment phase
Population: All enrolled and randomized participants were included in the endpoint analysis (ITT Population)
Measure: Mean (Standard Deviation); unit: Percentage of urine captured
Groups:
- PureWick System: PureWick™ System: The PureWick™ Female External Catheter (FEC) is intended for non-invasive urine output management in female patients. The PureWick™ FEC is a flexible, contoured external catheter that is positioned against the area where urine exits the female body. The PureWick™ FEC is connected to the PureWick™ Urine Collection System (PUCS) via connector tubing. The PUCS uses suction (not felt by the user) to pull voided urine through the device, regardless of the urine flow rate. Urine continues through vinyl tubing until it reaches a collection canister, away from the body.
- Hollister Female Urinary Pouch External Collection Device: Hollister® Female Urinary Pouch External Collection Device: The Hollister Female Urinary Pouch External Collection Device is intended to collect and contain urine for individuals with urinary incontinence. It is designed to be emptied and should be attached to a drainage bag. The FUP is made with hydrocolloid skin adhesive and polymer/copolymer plastics.
Arm/Group | PureWick System | Hollister Female Urinary Pouch External Collection Device
Number analyzed (Participants) | 11 | 5
Percentage of urine captured
  Overall | 79.3 (7.2) | 34.3 (18.5)
  Treatment Phase 1: number analyzed (Participants) | 6 | 3
  Treatment Phase 1 | 82.4 (6.0) | 24.2 (3.2)
  Treatment Phase 2: number analyzed (Participants) | 5 | 2
  Treatment Phase 2 | 75.6 (7.3) | 49.4 (24.2)
Statistical Analysis 1: Comparison: PureWick System vs Hollister Female Urinary Pouch External Collection Device; Test type: Superiority; p = 0.076, paired T-test; No formal hypothesis test was planned for this pilot study. P-values are provided for exploratory purposes and are unadjusted for multiplicity

2. Primary Outcome: Daily Average Skin Irritation Score Using the Draize Scale
Description: Draize Scale is a 5 point scale where 0 is no erythema, edema, or bleeding and 4 is severe erythema, edema, and/or bleeding.
  The primary safety endpoint of skin irritation score is derived by computing the mean of Draize Scale scores assessed daily during each study phase.
Time Frame: Daily for 28 days during each treatment phase
Population: All enrolled and randomized participants were included in the endpoint analysis (ITT Population)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PureWick System | Hollister Female Urinary Pouch External Collection Device
Number analyzed (Participants) | 11 | 5
score on a scale | 0.06 (0.12) | 0.03 (0.05)

3. Secondary Outcome: Nocturia Quality of Life (N-QOL) Score
Description: N-QOL is a standardized tool used to explore 13 items that might be affected by nocturia (e.g., concentration, productiveness, and low energy). Transformed Total Score is computed from the core 12 item summary scores and ranges from 0-100 with higher scores indicating better quality of life.
Time Frame: Starting at baseline and then every 2 weeks during each treatment phase
Population: All enrolled and randomized participants were included in the endpoint analysis (ITT Population). NQOL total scores were only analyzable for patients that missed up to 1 question. If more than 1 question was missed, total score could not be analyzed. Change in number analyzed over time is due to participant premature discontinuation.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PureWick System | Hollister Female Urinary Pouch External Collection Device
Number analyzed (Participants) | 11 | 5
score on a scale
  Baseline: number analyzed (Participants) | 11 | 4
  Baseline | 54.4 (25.8) | 55.7 (23.6)
  Week 1-2: number analyzed (Participants) | 9 | 2
  Week 1-2 | 60.0 (29.5) | 64.6 (2.9)
  Week 1-2 change from Baseline: number analyzed (Participants) | 9 | 2
  Week 1-2 change from Baseline | 6.7 (17.9) | 15.6 (25.0)
  Week 3-4: number analyzed (Participants) | 9 | 2
  Week 3-4 | 65.5 (23.1) | 47.9 (2.9)
  Week 3-4 change from Baseline: number analyzed (Participants) | 9 | 2
  Week 3-4 change from Baseline | 12.3 (15.4) | -1.0 (30.9)

4. Secondary Outcome: PROMIS Sleep Disturbance - Short Form 4a Score
Description: The PROMIS Sleep Disturbance Short Form 4a consists of 4 questions that each have 5 response options, with 1 indicating the least sleep disturbance and 5 indicating the most sleep disturbance. Total raw scores are translated into a T-score ranging from 32.0 to 73.3, with higher scores indicating worse outcome.
Time Frame: Starting at baseline and then every 7 days during each treatment phase
Population: All enrolled and randomized participants were included in the endpoint analysis (ITT Population). The PROMIS sleep disturbance questionnaire was added to the study in a protocol amendment; therefore, only one (1) participant was analyzed in each treatment group.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | PureWick System | Hollister Female Urinary Pouch External Collection Device
Number analyzed (Participants) | 1 | 1
score on a scale
  Baseline | 57.9 (3.3) | 54.3 (3.4)
  Day 8 | 52.4 (3.4) | 59.8 (3.3)
  Day 8 change from Baseline | -5.5 | 5.5
  Day 15 | 50.5 (3.4) | 56.1 (3.4)
  Day 15 change from Baseline | -7.4 | 1.8
  Day 22 | 54.3 (3.4) | 63.8 (3.4)
  Day 22 change from Baseline | -3.6 | 9.5
  Day 29 | 54.3 (3.4) | 57.9 (3.3)
  Day 29 change from Baseline | -3.6 | 3.6

5. Secondary Outcome: Participant's Tolerability of Device/Treatment
Description: Participant's tolerability is determined by the number of days of actual device use.
Time Frame: After completion of the 28-day treatment phase or at the time of treatment discontinuation, whichever comes first.
Population: All enrolled and randomized participants were included in the endpoint analysis (ITT Population)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | PureWick System | Hollister Female Urinary Pouch External Collection Device
Number analyzed (Participants) | 11 | 5
days
  Treatment Phase 1: number analyzed (Participants) | 6 | 3
  Treatment Phase 1 | 23.8 (9.3) | 10.7 (13.4)
  Treatment Phase 2: number analyzed (Participants) | 5 | 2
  Treatment Phase 2 | 23.2 (8.2) | 22.0 (7.1)

6. Secondary Outcome: Participant's Comfort Level Associated With Device/Treatment
Description: Overall comfort on a 5-point Likert scale ranging from 1- 5 with higher scores indicating a better outcome, where 1 = Very Uncomfortable, 2 = Uncomfortable, 3 = Neither Comfortable nor Uncomfortable, 4 = Comfortable, and 5 = Very Comfortable.
  The last question related to likelihood to recommend the device ranged from 1-5 with higher scores indicating a better outcome, where 1 = Very Unlikely, 2 = Unlikely, 3 = Neither Likely nor Unlikely, 4 = Likely, and 5 = Very Likely.
Time Frame: After completion of each 28-day treatment phase or at the time of treatment discontinuation, whichever comes first.
Population: All enrolled and randomized participants were included in the endpoint analysis (ITT Population)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PureWick System | Hollister Female Urinary Pouch External Collection Device
Number analyzed (Participants) | 11 | 5
score on a scale
  Comfort of Device Placement | 4.3 (0.7) | 2.5 (1.7)
  Comfort of Device During Sleep | 4.2 (1.0) | 3.0 (1.4)
  Comfort of Device Removal | 4.3 (0.5) | 1.0 (0.0)
  Likelihood to Recommend Device | 4.5 (1.0) | 1.0 (0.0)

7. Secondary Outcome: Participant's Opinion of Ease of Device Use
Description: Ease of use score on a 5-point Likert scale ranging from 1- 5 with higher scores indicating a better outcome, where 1 = Very Difficult, 2 = Somewhat Difficult, 3 = Average Difficulty, 4 = Somewhat Easy, and 5 = Very Easy.
  The last question related to dryness experienced with the device during sleep ranged from 1-4 with higher scores indicating a better outcome, where 1 = Never Dry, 2 = Sometimes Dry, 3 = Usually Dry, 4 = Always dry to mostly always dry
Time Frame: After completion of each 28-day treatment phase or at the time of treatment discontinuation, whichever comes first.
Population: All enrolled and randomized participants were included in the endpoint analysis (ITT Population)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PureWick System | Hollister Female Urinary Pouch External Collection Device
Number analyzed (Participants) | 11 | 5
score on a scale
  Ease of Device Placement | 4.4 (0.8) | 2.0 (0.8)
  Ease of Device Removal | 4.4 (0.8) | 2.0 (1.4)
  Dryness Experienced | 2.8 (1.1) | 1.3 (0.5)

ADVERSE EVENTS:
Time Frame: 28 days during each treatment phase
Arm/Group | PureWick System | Hollister Female Urinary Pouch External Collection Device
All-Cause Mortality (participants affected / at risk) | 0/11 | 1/5
Serious Adverse Events (participants affected / at risk) | 1/11 | 1/5
Other Adverse Events (participants affected / at risk) | 1/11 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PureWick System (N=11) | Hollister Female Urinary Pouch External Collection Device (N=5)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) — Participant was hospitalized for UTI
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Participant was hospitalized for dehydration
Death (General disorders) | 0 (0) | 1 (1) — Unknown cause of death
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PureWick System (N=11) | Hollister Female Urinary Pouch External Collection Device (N=5)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Rash - unknown cause
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-04-16): https://cdn.clinicaltrials.gov/large-docs/18/NCT05710718/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-11): https://cdn.clinicaltrials.gov/large-docs/18/NCT05710718/SAP_001.pdf